CLINICAL TRIAL: NCT05540964
Title: An Antiretroviral Treatment Interruption(ATI) Study to Evaluate the Impact and Durability of AGT103-T to Suppress Human Immunodeficiency Virus Replication in the Absence of Antiretroviral Therapy(ART) in Participants With Human Immunodeficiency Virus(HIV) Previously Treated With AGT103-T
Brief Title: An Antiretroviral Treatment Interruption (ATI) Study to Evaluate the Impact of Genetically Modified Autologous Cells (AGT103-T) to Suppress Human Immunodeficiency Virus Replication in the Absence of Antiretroviral Therapy
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: American Gene Technologies International Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: AGT-HC-169
Record Dates: First submitted 2022-09-08; First posted 2022-09-15 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-11

CONDITIONS: HIV
Keywords: Gene Therapy; Genetically modified CD4 T cells; Antiretroviral therapy interruption; Lentivirus vector

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single group: Study participants will be taken off antiretroviral therapy and blood samples will be collected during each clinic visit.
  Interventions: Other: Antiretroviral Therapy Interruption(ATI)

INTERVENTIONS:
Other: Antiretroviral Therapy Interruption(ATI) — Study participant that were previously infused with autologous genetically modified cell product will be taken off ART and followed closely by monitoring HIV rebound.

SUMMARY:
To test the hypothesis that AGT103-T cells therapy will allow HIV positive individual to reduce, modify or eliminate antiretroviral therapy.

DETAILED DESCRIPTION:
Study subjects who have been infused with AGT103-T in a prior trial (AGT-HC-168) will be invited to stop their antiretroviral therapy in two phases. The first antiretroviral interruption will be closely monitored and if at any point study termination criteria are met, the study participant will be placed back on antiretroviral therapy. The second antiretroviral therapy will be instituted once the inclusion criteria are met. The aim of two antiretroviral interruptions is to allow for adequate sensitization of the cells and expansion of the pool of infused gene-modified cells. The two-phased ATI allows for a more robust suppression of HIV in study participants. Participants are monitored closely to determine if the autologous T cells with which they were previously infused, modify the kinetics of HIV rebound. The study participant will be closely monitored for the recurrence of HIV viremia and a decrease in their CD4 lymphocyte number.

ELIGIBILITY:
Inclusion Criteria:

1. Successful engraftment of AGT103-T with at least 30 days post-infusion safety monitoring during the AGT-HC-168 Parent Study.

   Note: Successful engraftment is defined as detectable levels of AGT103-T cells bearing the AGT103 lentivirus vector.
2. HIV <50 copies of viral RNA/mL plasma on stable ART.
3. Continuation on the same ART regimen during the AGT-HC-168 Parent Study unless change in treatment with ART regimen is medically indicated.
4. CD4 T cell count >400 cells/mm3.
5. Ability to understand the study and willingness to comply with study-required procedures and visits.
6. Written informed consent signed and dated by the study participant.
7. A negative pregnancy test for females of childbearing potential. A female participant is considered to be of childbearing potential if she is menstruating, has an intact uterus and at least 1 ovary, and is less than 2 years postmenopausal.
8. Unless medically prescribed, a negative drug test for amphetamines; barbiturates; benzodiazepines; cocaine; methadone (Dolophine®); opiates (codeine, morphine only); phencyclidine (PCP); propoxyphene.
9. Female participants of childbearing potential and male participants who are sexually active with a partner of childbearing potential must agree to use an adequate method of contraception at screening and throughout trial participation.
10. Female and male participants who are sexually active with a partner must agree to abstain from sexual activity or use an adequate method of protection (e.g., condoms) at screening and throughout trial participation.
11. Agree to not receive immunosuppressive and/or investigational therapies during the study.

    Note: Prohibited immunosuppressive medications do not include corticosteroid nasal spray or inhaler; topical corticosteroids for mild, uncomplicated dermatitis; or oral/parenteral corticosteroids given for non-chronic conditions.
12. Has adequate organ function as indicated by the following laboratory values:

    * Hematocrit ≥33% or hemoglobin ≥13 g/dL (males) and ≥12 g/dL (females)
    * Platelet count ≥150,000/mm3
    * Absolute neutrophil count ≥1,500/mm3
    * Serum creatinine ≤1.3 times ULN or calculated creatinine clearance (for those with creatinine >1.3 ULN) ≥60 mL/min
    * Prothrombin Time or INR ≤ 1.5 times ULN
    * Total bilirubin <1.5 times the ULN range. If total bilirubin is elevated, direct bilirubin must be < 2 times the ULN range, except in participants with Gilbert's Syndrome who must have serum bilirubin <3.0 times ULN (NOTE: If participant is on an atazanavir containing therapy then a direct bilirubin should be measured instead of the total bilirubin and must be ≤ 1.0 mg/dL. Also, asymptomatic elevations due to ART medications are not exclusionary when, in the opinion of the Investigator, the abnormalities are not attributable to intrinsic hepatic disease.
    * Amylase < 3.0 times ULN at the time of screening
    * AST (SGOT) and ALT (SGPT): ≤ 3.0 times ULN

Exclusion Criteria

1. Any Grade 3 or higher drug product-related AE in the AGT-HC-168 Parent Study (participant may be enrolled once AE resolved).
2. Any change in health status that would exclude enrollment in the AGT-HC-168 Parent Study.
3. Active viral hepatitis B or hepatitis C infection. A complete hepatitis B virus (HBV) screen (B core antibody, HBV surface antibody, and HBV surface antigen testing) must be completed. Viral load testing will be used in questionable cases, per the discretion of the Investigator.

   * The results for hepatitis B may be positive for surface antibodies against HBV but must be negative for circulating HBV surface antigen to confirm the absence of active infection.
   * The results for hepatitis C virus (HCV) may be positive for antibodies against HCV but must be negative for HCV viral RNA in blood to confirm the absence of active infection.
4. History of or current cancer or malignancy, with the exception of successfully treated basal cell carcinoma of the skin.
5. Current diagnosis of New York Heart Association Grade 3 or 4 congestive heart failure, uncontrolled angina, or arrhythmias.
6. Any clinically significant renal, hepatic, or pulmonary disease.
7. Is being treated for culture-confirmed bacteremia or had culture-confirmed bacteremia within 1 month prior to screening.
8. Has signs or symptoms of acute infectious disease.
9. Significant laboratory values and/or chronic medical condition that in the opinion of the Principal Investigator could impact trial participation.
10. Currently pregnant or breast-feeding.
11. Unwilling to use acceptable methods of birth control from the time of study entry to 1 month after restart of ART if sexually active with opposite sex. The following are acceptable methods of birth control: condoms (male or female) with or without a spermicidal agent, intrauterine device, diaphragm or cervical cap with spermicide, or hormonal-based contraception.
12. Active alcohol use or dependence that, in the opinion of the Investigator, would interfere with adherence to study requirements.
13. Serious illness requiring systemic treatment and/or hospitalization within 30 days prior to screening.
14. Subject is unwilling to agree to practice safe sex or share needles.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subject who were infused with the investigational product AGT103-T in the AGT168 clinical trial
Sampling Method: Probability Sample
Enrollment: 7 (Estimated)
Dates: Start 2022-07-19 (Actual); Primary Completion 2025-07-19 (Estimated); Study Completion 2025-07-19 (Estimated)

PRIMARY OUTCOMES:
HIV kinetics | 3 Years
  Observe for changes in the HIV viral load.
CD T cell changes | 3year
  Observe the changes in the CD4 T cells and CD8 T cells count following antiretroviral treatment interruption(ATI)

SECONDARY OUTCOMES:
Assess the durability of AGT103-T gene-modified cells during and after ATI | 3 Year
  Measure the AGT103-T gene-modified cell during and after ATI
CD T cells changes | 3 Years
  Measure changes in frequency of Gag-specific CD4 and CD8 T cells following ATI

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Georgetown University, Washington D.C., District of Columbia
  - Washington Health Institute, Washington D.C., District of Columbia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Jain A, Liou ML, Xiao L, Canepa GE. Impact of AGT103-T cell and gene therapy on intact HIV proviral reservoirs. AIDS. 2026 Feb 11. doi: 10.1097/QAD.0000000000004459. Online ahead of print. PMID 41670418